CLINICAL TRIAL: NCT04158505
Title: Real World Study on the Efficacy and Safety of Pyrotinib in the Treatment of HER2 Positive Breast Cancer: An Observational,Multi-center,Prospective Study (Real Pretty Study)
Brief Title: Real World Study of Pyrotinib in Human Epidermal Growth Factor Receptor-2 (HER2) Positive Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Binghe Xu, chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: HR-BLTN-016
Record Dates: First submitted 2019-11-07; First posted 2019-11-08 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: HER2-positive Breast Cancer
Keywords: pyrotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- non-interventional study
  Interventions: Other: non-interventional

INTERVENTIONS:
Other: non-interventional — This prospective, observational study will be conducted according to each site's routine clinical practice

SUMMARY:
This Non-Interventional Study will describe and analyze the clinical use of pyrotinib in clinical practice in the treatment of HER2 positive breast cancer in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old with histologically confirmed HER2 positive breast cancer.
2. Documented HER2 overexpression by local laboratory ,defined as immunohistochemistry (IHC) 3+ or fluorescence in situ hybridization (FISH) positive.
3. Physician has determined that treatment with pyrotinib is indicated.
4. Traceable medical record available.

Exclusion Criteria:

1. Patients who are unable to understand the nature of the study and are unwilling to sign an informed consent .
2. Pregnant or breast feeding patients
3. Patients participating in any interventional clinical trial that includes investigational or marketed products at the time of enrollment.
4. Patients not suitable for this study under investigators' consideration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2+ breast cancer patients whose treatment decision with pyrotinib has been made by their physician and who meet the eligibility criteria will be invited to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | 12 months
  Progression Free Survival(PFS)
Pathological Complete Response（pCR）Rate | through study completion, an average of 1 year
  Percentage of Participants With Pathological Complete Response
Incidences of adverse events and toxicities | through study completion, an average of 1 year
  Incidences of adverse events and toxicities

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Cancer Hospital/Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided